CLINICAL TRIAL: NCT00209495
Title: Effect of Paracetamol Versus Paracetamol Combined With Pregabalin Versus Paracetamol Combined With Pregabalin and Dexamethasone on Pain and Opioid Requirements in Patients Scheduled for Abdominal Hysterectomy.
Brief Title: Effect of Paracetamol,Pregabalin and Dexamethasone on Pain and Opioid Requirements in Postoperative Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: SM1-04
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2008-02-29 (Estimated); Status verified 2008-02

CONDITIONS: Pain, Postoperative
Keywords: Abdominal hysterectomy; Pregabalin; Dexamethasone; Multimodal postoperative analgesia
MeSH Terms: conditions — Pain, Postoperative | interventions — Pregabalin; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A (Placebo Comparator)
  Interventions: Drug: Pregabalin; Dexamethasone
- B (Experimental): Pregabalin
  Interventions: Drug: Pregabalin; Dexamethasone
- C (Experimental): Pregabalin + dexamethasone
  Interventions: Drug: Pregabalin; Dexamethasone

INTERVENTIONS:
Drug: Pregabalin; Dexamethasone — Comparing combinations of paracetamol + pregabalin 300 mg + dexamethasone 8 mg

SUMMARY:
Women scheduled for abdominal hysterectomy needs postoperative pain treatment, i.e. morphine. Unfortunately morphine has side-effect: nausea, vomiting, sedation and dizziness, which is unpleasant for the patients and sometimes keeps them at bed longer time than needed. We investigate in new combinations of analgesics for postoperative pain, hoping to minimize the need for morphine.

DETAILED DESCRIPTION:
Combinations of paracetamol versus paracetamol + pregabalin versus paracetamol + pregabalin + dexamethasone is investigated. Primary outcome is 24 hours morphine usage.

ELIGIBILITY:
Inclusion Criteria:

* Women scheduled for abdominal hysterectomy, between the age of 18 and 75, ASA 1-2
* BMI between 18-32.

Exclusion Criteria:

Patients who:

* Are unable to cooperate
* Has cancer ovarian
* Does not speak Danish
* Has allergy for drugs used in the trial
* Has drug and medicine abuse
* Epilepsy
* Diabetes treated with medicine
* Chronic pain condition
* Daily use of antacids or analgesic
* Known kidney disease
* Use of antidepressive

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2005-06; Primary Completion 2007-11 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
The total amount of morphine needed postoperatively form 0 - 4 h, and 0 - 24 h, administered by the patient controlled pain treatment. (PCA) | 0 - 24h

SECONDARY OUTCOMES:
Pain Score (VAS) at rest and at mobilisation. | 0 - 24h
Postoperative nausea and vomiting. | 0 - 24h
Sedation. | 0 - 24h
Dizziness. | 0 - 24h
All measurements are taken at 2, 4 and 24 h postoperatively. | 0 - 24h

CONTACTS AND LOCATIONS:
Overall Officials: Ole Mathiesen, MD, Principal Investigator — Department of Anaesthesiology, Copenhagen University Hospital in Glostrup, 2600 Glostrup, Denmark
Locations (2):
- Denmark (2):
  - Operations og Anæstesiologisk afd. Y, KAS Glostrup, Glostrup Municipality, Copenhagen
  - Herning Centralsygehus, Herning